CLINICAL TRIAL: NCT04065646
Title: Nutrition Ed, Access and Texting (NEAT): Combining the Hartford Mobile Market With e-Marketing
Brief Title: Nutrition Education and e-Texting to Increase Access to Fresh Produce
Acronym: (NEAT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sofia Segura-Pérez (Other)
Collaborators: Yale University (Other); Cornell University (Other)
Responsible Party: Sponsor-Investigator, Sofia Segura-Pérez, Associate Nutrition Unit Director, Hispanic Health Council, Inc.
Organization: Hispanic Health Council, Inc. (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HHCNEAT2015
Record Dates: First submitted 2019-08-02; First posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Healthy Eating
Keywords: Food Access; Food Security; Fruits and Vegetables; Low-Income

STUDY DESIGN:
Intervention Model Description: Baseline interviews will be conducted after participation in nutrition education activity. Upon completing baseline, participants will be randomized into intervention (HMM text messaging) or control (non-health-related texting) groups. Texting will begin the day after randomization is completed and will occur once daily during business days for a duration of one month. In addition to HMM access messages, intervention group participants will receive texts with links to four $5.00 incentive coupons for the Hartford Mobile Market, one during each of the four weeks that the texting will take place. Follow-up interviews will be conducted two weeks after the end of the one-month texting period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive daily text messages with information on: (i) HMM stop locations and schedule; (ii) information on HMM weekly produce specials and sales; (iii) motivational messages encouraging use of the HMM; and (iv) links to produce coupons that they can exchange at HMM- $5 coupons received weekly for the four-week texting period.
  Interventions: Other: Mobile
- Control (No Intervention): The control group will receive the same dosage of daily text messages covering free activities taking place at the Hartford Public Library and other community locations. The control group will not receive incentive coupons.

INTERVENTIONS:
Other: Mobile
  Arms: Intervention

SUMMARY:
The proposed project, Nutrition Ed, Access and Texting (NEAT): Combining the Hartford Mobile Market with e-Marketing , uses an e-technology social marketing strategy to promote use of a recently launched mobile produce market among SNAP-Ed recipients. This study will potentially increase fresh produce access and intake by combining an innovative food system change (produce mobile market) with existing SNAP-Ed nutrition education curriculum and the use of e-marketing technology.

DETAILED DESCRIPTION:
The proposed project, Nutrition Ed, Access and Texting (NEAT): Combining the Hartford Mobile Market with e-Marketing uses an e-technology social marketing strategy to promote use of a recently launched mobile produce market among SNAP-Ed recipients. This study will potentially increase fresh produce access and intake by combining an innovative food system change (produce mobile market) with existing SNAP-Ed nutrition education curriculum and the use of e-marketing technology. Thus, the study combines key elements that have been deemed necessary for increasing produce intake among low income communities. The goal of the NEAT study is to assess the impact of a texting-based social marketing campaign on SNAP-Ed participants' access to and purchase of fresh produce on a recently launched mobile produce market, and their subsequent produce intake. Objectives include: 1) Compare the impact of nutrition education alone to nutrition education plus promotional text messaging on purchase of fruits and vegetables; 2) Compare the impact of nutrition education alone to nutrition education plus promotional text messaging on consumption of fruits and vegetables; and 3) Assess the effectiveness of coupon distribution on coupon redemption at a mobile produce market. The NEAT design will be a randomized controlled trial using a pre-post assessment comparing change in behavior. Both intervention and control groups will receive SNAP-Ed education as currently delivered by the Hispanic Health Council. The intervention group will receive additional promotional text messaging related to use of the mobile market. The control group will receive text messaging about free activities taking place at the Hartford Public Library and other community locations. Participants will be interviewed via phone at baseline, then randomized to intervention and control groups, and re-interviewed again 6 weeks after they start receiving the text messages, which it will be 2 weeks after the one-month texting period ends.

ELIGIBILITY:
Inclusion Criteria:

* SNAP eligible participants with children under 5 years old living at home.
* Living in Hartford, CT.
* Having a cell phone with unlimited smart phone data plans.

Exclusion Criteria:

* Not living in Hartford Less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-10-23 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Change in consumption of fruits | Baseline and 6 weeks follow up
  Measured with one question about daily consumption of fruits from a seven item fruit and vegetable checklist developed by Townsend et.al.
Change in consumption of vegetables. | Baseline and 6 weeks follow up
  Measured with a one question from a seven item fruit and vegetable checklist developed by Townsend et.al.
Change in fruits eating behaviors Increase consumption of fruits and vegetables | Baseline and 6 weeks follow up
  Measured with a readiness 5 item continuous scale item for fruits from fruit and vegetable inventory validated by Townsend et.al.
Change in vegetables eating behaviors. Increase consumption of fruits and vegetables | Baseline and 6 weeks follow up
  Measured with a 5 item continuous scale from vegetables from fruit and vegetable inventory validated by Townsend et.al.
Change in amount of money spent on fruits and vegetables. | Baseline and at 6 week follow up
  self-reported amount of money spent on fresh produce per month.
Change in amount of money spent on fruits. | Baseline and at 6 week follow up
  self-reported amount of money spent on fruit per week.
Change in amount of money spent on vegetables. | Baseline and at 6 week follow up
  self-reported amount of money spent on vegetables per week.
Change in self reported usage of the Hartford Mobile Market for buying fresh produce | baseline and at 6 weeks follow up
  self-reported participant's usage of mobile market (yes/no)

SECONDARY OUTCOMES:
Participant utilization of coupons | 6 week follow up
  Based on one yes/no question about coupon redemption
Participant's satisfaction with e-texting messages (likeness) | 6 weeks follow up
  Self reported satisfaction with nutrition messages using a 5- likert scale (like it very much to dislike it very much)
Participant's assessment of usefulness of the messages | 6 weeks follow up
  Self reported continuous 4 likert scale from not useful to very much useful.
Participant's assessment of usefulness of the coupons | 6 week follow up
  Self reported continuous 4 likert scale from not useful to very much useful.

IPD SHARING:
Plan to Share IPD: No